CLINICAL TRIAL: NCT04772898
Title: Effectiveness of a 6-week Hippotherapy Program in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Anastasia Kyvelidou, Assistant Professor, Creighton University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5R03HD101115-02 (NIH)
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Autism Spectrum Disorders (Experimental): Children with autism spectrum disorder will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Interventions: Behavioral: Hippotherapy
- Children with typical development (Active Comparator): Children with autism spectrum disorder and with typical development will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Interventions: Behavioral: Hippotherapy

INTERVENTIONS:
Behavioral: Hippotherapy — The hippotherapy involves occupational therapy while being on a horse.

SUMMARY:
The prevalence of autism spectrum disorders (ASD) has increased dramatically in the last decade. The increasing occurrence of ASD creates an imperative need to test the effectiveness and efficacy mechanisms of appropriate interventions. Hippotherapy (HPOT) is a treatment option that has been show beneficial for children with ASD as well as other children with developmental disorders. The current projects focuses on understanding the mechanisms of HPOT efficacy and evaluating a short-term HPOT program for children with ASD.

DETAILED DESCRIPTION:
The incidence of autism spectrum disorders (ASD) has increased dramatically in the last decade. The latest report from the Centers for Disease Control and Prevention state that 1 in 59 children are being diagnosed with ASD and it is four times more prevalent in boys than girls. Common treatments for children with ASD are applied behavioral therapy, occupational and speech therapy, which are used solely or in combination. Hippotherapy (HPOT) is another treatment option that has been shown to positively impact various aspects of behavior. This pilot project aims to determine the effects of a 6-week HPOT program on movement and social behavior of children with ASD and to investigate the underlying mechanisms of why HPOT is successful for ASD through the coupling of physiological and temperamental responses between horse and rider. The approach involves examining these skills pre, during, and post HPOT intervention in children diagnosed with ASD. A group of aged matched children with typical development will serve as the control group. Innovative measures of physiological coupling and temperament between horse and rider as well as objective and quantitative measures of movement and social behavior and caregiver perception will be collected. The investigators anticipate that following completion of the proposed study, they will provide the necessary foundation to understand the mechanisms of HPOT, and thus provide a new framework to test clinical trials of HPOT and human-animal interaction, and ultimately improve the lives of those diagnosed with ASD and their families.

ELIGIBILITY:
For the children with Autism Spectrum Disorders:

Inclusion Criteria:

1. diagnosis of ASD based upon the Autism Diagnostic Observation Schedule and parent interview,
2. medical approval for participation in the HPOT activity,
3. no other medical or psychiatric diagnoses besides ASD
4. tolerate helmet on head and attachments of the movement and heart rate sensors.

The inclusion criteria for the TD children will be:

1. no diagnosis or family history of ASD
2. no other neurodevelopmental or musculoskeletal disorder
3. tolerate helmet on head and attachments of the movement and heart rate sensors.
4. medical approval for participation in the HPOT activity,

Exclusion Criteria:

1. under 5 years of age or over 10 years of age
2. has a serious comorbid medical diagnosis
3. major vision or hearing impairments
4. severe behavioral problems
5. an orthopedic or genetic diagnosis

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Kyvelidou, PhD, Principal Investigator — Creighton University
Locations (1):
- Hearthland Equine Therapeutic Riding Academy, Gretna, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events
Groups:
- Children With Autism Spectrum Disorder: Children with autism spectrum disorder will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Hippotherapy: The hippotherapy involves occupational therapy while being on a horse.
- Children With Typical Development: Children with typical development will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Hippotherapy: The hippotherapy involves occupational therapy while being on a horse.
Period: Overall Study
Arm/Group | Children With Autism Spectrum Disorder | Children With Typical Development
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Autism Spectrum Disorders | Children With Typical Development | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8 (1.97) | 7.8 (1.44) | 7.9 (1.715)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 15 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Social Responsiveness Scale (SRS) [Mean (Standard Deviation); unit: Points] — Population: One child from the typical development group dropped out, so we did not include them in the analysis
  Points
    number analyzed (Participants) | 15 | 14 | 29
    (all) | 16.5 (12.4) | 89.06 (27.3) | 52.78 (19.85)

OUTCOME MEASURES:

1. Primary Outcome: Social Responsiveness Scale (SRS)
Description: The SRS provides a clear picture of a child's social impairments, assessing social awareness, social information processing, capacity for reciprocal social communication, social anxiety/avoidance, and autistic preoccupations and traits. The SRS is a 65-item rating scale that measures autism traits over the previous 6 months in children and adolescents aged 4-18 years. Each item is scaled from 0 (never true) to 3 (almost always true), generating a total score ranging from 0 to 195.The total score of the SRS is reported below. Higher values represent worse outcome.
Time Frame: Change from Pre (baseline) to Post (after completion of 6 weeks of intervention)
Population: Children with typical development and diagnosed with ASD based on the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Children With Typical Development | Children With Autism Spectrum Disorder
Number analyzed (Participants) | 14 | 15
Points
  Pre | 16.5 (12.4) | 89.06 (27.3)
  Post | 14.5 (12.3) | 79.8 (29.5)

2. Primary Outcome: Postural Control
Description: Postural control assessment with a force platform with eyes open and eyes closed. Differences were more prevalent with eyes closed. We report a specific measure of postural control which is median frequency while standing with eyes closed. Median frequency can have a very wide range of values, but increased values of median frequency suggest faster postural control adaptations.
Time Frame: Change from Pre (baseline) to Post (6 weeks after hippotherapy intervention)
Population: The standing postural control protocol required children to be able to stand with eyes open and closed for 10 sec without moving their legs. This was possible only for 8 children with the autism spectrum disorder group and all of the children in the typical development group.
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Children With Typical Development | Children With Autism Spectrum Disorder
Number analyzed (Participants) | 14 | 8
Hz
  Pre | 0.525 (0.17) | 0.48 (0.18)
  Post | 0.53 (0.21) | 0.57 (0.15)

3. Primary Outcome: Cross Sample Entropy Between the Heart Rate Sensors of the Horse and Rider
Description: Heart rate monitors were placed around the upper thorax of both the rider and horse and simultaneously began collecting data at the beginning of each session. Data was collected at the first, third, and sixth sessions of the intervention. We used the heart rate signals of the horse and rider to calculate the Cross approximate entropy. Cross-ApEn quantifies the regularity of patterns in a pair of related time series and is indicative of the dimensionality of control of the two signals. The calculation of Cross-ApEn is similar to approximate entropy with the exception that successive two-point vectors of one signal are compared with current and previous two-point vectors of another signal. Larger Cross-ApEn values indicate greater joint signal asynchrony while lower Cross-ApEn values indicate greater joint signal synchrony.For details on calculation of Cross-ApEn please refer to: Pincus S, Singer BH. Randomness and degrees of irregularity. Proc Natl Acad Sci USA. 1996; 93: 2083-2088.
Time Frame: During week 1, week 3 and week 6 of the treatment sessions
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Children With Autism Spectrum Disorder | Children With Typical Development
Number analyzed (Participants) | 15 | 14
Unitless
  1st session | 0.685 (0.09) | 0.512 (0.25)
  3rd session | 0.644 (0.18) | 0.578 (0.16)
  6th session | 0.681 (0.18) | 0.564 (0.18)

4. Secondary Outcome: Correlation Between Horse Temperament and Therapeutic Outcomes
Description: Correlation estimate between horse temperament and treatment effectiveness
Time Frame: from baseline to 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Aberrant Behavior Checklist
Description: This is a questionnaire completed by the caregivers that assesses irritability, social withdrawal, stereotypic behavior, hyperactive/noncompliance, inappropriate speech
Time Frame: Change from baseline to 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the intervention and participation to the study which was 8 weeks.
Groups:
- Children With Typical Development: Children with typical will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Hippotherapy: The hippotherapy involves occupational therapy while being on a horse.
- Children With Autism Spectrum: Children with autism spectrum disorder will receive a 6 week (once per week) hippotherapy protocol. During the hippotherapy session, the researchers will monitor the heart rate variability of the horse and the rider. Both horse and rider will wear an electrode strap around the upper thorax. Heart rate recordings will be started simultaneously at the beginning of the HPOT session. To assess movement coupling between the horse and rider, five tri-axial inertial sensors (OPAL, APDM, Inc, Portland, OR) will be used. The sensors will collect actively synchronized tri-axial accelerometer and gyroscope data. One inertial sensor will be placed dorsal at the rider's pelvis, one frontal at the top of the forehead, and one frontal at the top of the sternum. The sensors on the horse will be fixed on the back of the horse on the spine level between T8 and T10 and on the head.
  Hippotherapy: The hippotherapy involves occupational therapy while being on a horse.
Arm/Group | Children With Typical Development | Children With Autism Spectrum
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04772898/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04772898/ICF_001.pdf